CLINICAL TRIAL: NCT03124901
Title: Accuracy of Noninvasive Pulse Oximeter Measurement of Hemoglobin for Rainbow DCI Sensor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TR-17636-56044
Record Dates: First submitted 2017-04-11; First posted 2017-04-24 (Actual); Results first posted 2017-06-12 (Actual); Last update posted 2017-06-12 (Actual); Status verified 2017-05

CONDITIONS: Surgery; Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Test Group (Experimental): All subjects are enrolled into the test group and all subjects receive DCI pulse oximeter sensor.
  Interventions: Device: DCI pulse oximeter sensor

INTERVENTIONS:
Device: DCI pulse oximeter sensor

SUMMARY:
In this study, the concentration of hemoglobin within the subject's blood is affected by fluid status changes. The fluid status is affected by fluid loss during surgery for hospitalized study subjects or controlled administration of fluids intravenously for healthy study volunteers. The accuracy of a noninvasive hemoglobin sensor(s) will be assessed by comparing with blood sample analysis.

ELIGIBILITY:
Inclusion Criteria:

* Has physical status between ASA 1 or 2
* Able to communicate in English

Exclusion Criteria:

* Pregnant or sexually active without birth control.
* Hemoglobin less than 11g/dL
* Known alcohol or drug abuse
* Skin abnormalities affecting the digits such as psoriasis, eczema, angioma, scar tissue, burn, fungal infection
* Nail polish
* Head injury with loss of consciousness within the last year
* Known neurological and psychiatric conditions.
* Known concurrent chronic usage of psychoactive or anti-convulsive drugs within the last 90 days, or use in the last 7 days (i.e. tricyclic antidepressants, MAO inhibitors, lithium, neuroleptics, anxiolytics or antipsychotics. Except SSRIs
* Subject has any medical condition which, in the judgement of the investigator, renders them inappropriate for participation in this study, such as Reynods syndrome
* Hypertension: Systolic BP >= 140 mmHg or Diastolic BP >= 90 mmHg
* Baseline heart rate <50 beats per minute

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2008-09-30 (Actual); Primary Completion 2008-10-27 (Actual); Study Completion 2008-10-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Masimo Clinical Lab, Irvine, California
  - Loma Linda University Medical Center, Loma Linda, California

RESULTS

PARTICIPANT FLOW:
Groups:
- Test Group: All subject are enrolled into the test group and all subjects receive DCI pulse oximeter sensor.
Period: Overall Study
Arm/Group | Test Group
Started | 147
Completed | 147
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Test Group
Number analyzed (Participants) | 147
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 147
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43
  Male | 104
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 147

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of Sensor
Description: Accuracy willl be determined by comparing the noninvasive hemoglobin measurement of the pulse oximeter to the hemoglobin value obtained from a blood sample and calculating the arithmetic root mean square(Arms) error value.
Time Frame: Up to 24 hours
Measure: Number; unit: g/dL
Arm/Group | Test Group
Number analyzed (Participants) | 147
g/dL | 0.98

ADVERSE EVENTS:
Arm/Group | Test Group
All-Cause Mortality (participants affected / at risk) | 0/147
Serious Adverse Events (participants affected / at risk) | 0/147
Other Adverse Events (participants affected / at risk) | 0/147

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less